CLINICAL TRIAL: NCT07351006
Title: Exercise as Medicine: A Non-Pharmacological Approach to Menopausal Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linnaeus University (Other)
Responsible Party: Principal Investigator, Sofia Ryman Ryman Augustsson, Associate Professor, Linnaeus University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-06613-01
Record Dates: First submitted 2025-12-16; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Menopause Syndrome; Sleep Disturbance
MeSH Terms: conditions — Parasomnias | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to 1) Intervention with strength training (n=15); 2) Intervention with dance-based training (n=15) or 3) control group (n=15).
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessors are blinded to the type of intervention (or control) that the participants are assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Strength training (Experimental): Strength training intervention.
  Interventions: Other: Strength training
- Dance-based training (Experimental): Dance-based training intervention.
  Interventions: Other: Dance-based training
- Control (No Intervention): No intervention

INTERVENTIONS:
Other: Strength training — The strength training intervention consists of an 8-week program performed 3 times per week, with sessions lasting ~30 minutes. Designed by a licensed physiotherapist, the program targets major muscle groups and includes a warm-up followed by structured exercises.
  Training uses body weight and simple household equipment, such as chairs and filled water bottles, at an intensity of 8-12 repetition maximum. Each exercise has three to four difficulty levels. Before starting, participants test and select an appropriate level for each exercise to ensure correct intensity.
  Participants perform at a level allowing at least eight repetitions and progress once they can complete more than twelve. This enables individualized, progressive training. After each session, participants record the difficulty level and number of repetitions in a training diary. For the full-scale intervention, exercise selection, intensity, and volume may be adjusted, and the program will be extended to 15 weeks.
  Arms: Strength training
Other: Dance-based training — Participants in the dance-based intervention will exercise three times per week at moderate intensity, following a structured 30-minute program performed individually at home via pre-recorded sessions.
  After each session, participants will complete a training diary and rate perceived exertion using the Borg RPE scale (6-20), targeting at least moderate intensity (RPE ≥ 14), adjusting effort accordingly.
  The program was developed and recorded by a licensed physiotherapist, pilot-tested with a small group, and reviewed by a supervising expert who provided feedback. Participants can ask questions and receive guidance on performing the exercises.
  For the full-scale intervention, exercise selection, intensity, and volume may be refined, and the program will be conducted over 15 weeks.
  Arms: Dance-based training

SUMMARY:
The aim of this clinical trial is to evaluate the effects of different forms of physical exercise in women experiencing menopausal symptoms. Specifically, the project investigates the effects of: (1) strength training on women's perceived menopausal symptoms; (2) dance-based exercise on women's perceived menopausal symptoms; and (3) adherence to structured, digital home-based exercise programs.

The following research questions will be addressed within the framework of the project:

Does regular strength training reduce women's perceived menopausal symptoms?

To what extent does strength training influence menopausal symptoms and sleep quality in women?

What is the level of adherence to a digital, home-based strength training program among women with menopausal symptoms?

Does regular dance-based physical activity reduce women's perceived menopausal symptoms?

To what extent does dance-based physical activity influence menopausal symptoms and sleep quality in women?

What is the level of adherence to a digital, home-based dance exercise program among women with menopausal symptoms?

Which exercise protocol-strength training or dance-based exercise-has the greatest effect on perceived menopausal symptoms?

The researchers will compare a digital, home-based strength training program with a digital, home-based dance exercise program, as well as with a control group, to determine which type of exercise has the greatest effect on menopausal symptoms and sleep quality.

Participants will:

Perform either dance-based exercise or strength training for 8 weeks, three times per week, following a structured program of approximately 30 minutes per session, or participate as part of the control group.

Complete validated questionnaires assessing menopausal health, including somatic, psychological, and sexual symptoms, as well as perceived quality of life and sleep quality, both before and after the intervention.

Maintain a training diary to monitor adherence and progression, including increases in training intensity

DETAILED DESCRIPTION:
This clinical trial will be conducted as a randomized controlled trial, in which participants will be randomly assigned to either an intervention group or a control group. The study will begin with a pilot phase including 45 menopausal women, who will be randomly allocated to one of three groups: (1) strength training intervention (n = 15); (2) dance-based training intervention (n = 15); or (3) control group (n = 15).

Following completion of the pilot study, a full-scale intervention trial will be conducted. The sample size for the main study will be determined by a power calculation based on the results obtained from the pilot phase.

The study will begin with an assessment of participants' menopausal health, including somatic, psychological, and sexual symptoms, as well as perceived quality of life and sleep quality. These outcomes will be measured using the Menopause Rating Scale (MRS) and the Pittsburgh Sleep Quality Index (PSQI).The training protocols will be conducted over an 8-week period, with sessions performed three times per week according to a structured program lasting approximately 30 minutes per session. Two weeks after completion of the intervention, participants will be reassessed using the same instruments, with questionnaires distributed electronically via SurveyMonkey®.

The intervention will begin with a digital introductory meeting, during which participants will receive information materials on menopausal symptoms and a detailed review of the training program and study procedures. Participants in the control group will continue their usual daily activities without any prescribed intervention throughout the 8-week study period. Participants in the control group will be assessed using both instruments on two occasions, with an 8-week interval between assessments. Upon completion of the study, control group participants will be offered access to both intervention programs, as well as the results from Studies 1 and 2.

Throughout the study period, participants will be instructed not to introduce any additional forms of exercise or make changes to existing physical activity habits. The full-scale intervention is planned to be conducted over a 15-week period with a potentially larger sample size.

ELIGIBILITY:
Inclusion Criteria:

* Biological female sex
* Age 45-55 years
* Experiencing menopausal symptoms, defined as irregular or altered menstruation plus at least one of the following:
* Hot flashes or sweating
* Sleep problems
* Mood swings or depression
* Dry mucous membranes
* Recurrent urinary tract infections or overactive bladder
* Joint pain
* Decreased libido
* Weight gain

Exclusion Criteria:

* Have taken medication or natural remedies for menopausal symptoms in the past 2 months
* Menopause due to illness or surgical intervention
* Medical conditions that contraindicate participation in the exercise intervention
* Engaged in physical activity for ≥150 minutes per week, including ≥ 75 minutes at high intensity

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Menopause Rating Scale (MRS) | 2 times: 1) Baseline: Day 1 and 2) Post intervention: week 8
  The Menopause Rating Scale (MRS) consists of 11 items grouped into three dimensions:
  * Somatic Symptoms: Hot flashes, joint pain, and related physical complaints.
  * Psychological Symptoms: Depressive mood, irritability, anxiety, and similar issues.
  * Urogenital Symptoms: Bladder problems, vaginal dryness, and related concerns. Each item is rated on a 5-point Likert scale from 0 (not present) to 4 (very severe). The total score, calculated by summing all items, provides an overall measure of menopausal symptom severity. Thus, total score ranging from 0-44.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | 2 times: 1) Baseline: Day 1 and 2) Post intervention: week 8
  Sleep quality is assessed using the Pittsburgh Sleep Quality Index (PSQI), which evaluates seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Each component is scored from 0 to 3, and a global score is calculated by summing the components. Higher scores indicate poorer sleep quality. The Pittsburgh Sleep Quality Index (PSQI) generates a global score ranging from 0 to 21, where a score greater than 5 typically indicates poor sleep quality. This threshold serves as a clinical benchmark, with higher scores correlating with increased severity of sleep disturbances.

CONTACTS AND LOCATIONS:
Locations (1):
- Sofia Ryman Augustsson, Kalmar, Sweden

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-11-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT07351006/SAP_000.pdf